CLINICAL TRIAL: NCT01553877
Title: Development and Acceptability Testing of Ready-to-use-complementary Food Supplement (RUCFS) for Children in Bangladesh
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PR-10066
Record Dates: First submitted 2012-01-24; First posted 2012-03-14 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-03

CONDITIONS: Moderately Malnourished Children
MeSH Terms: interventions — Molasses; Soybean Oil

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pushti Packet (Active Comparator)
  Interventions: Dietary Supplement: Pushti packet
- Rice based Ready to Use Complementary Food Supplements (Experimental)
  Interventions: Dietary Supplement: Rice based Ready to Use Complementary Food Supplements
- Chick-pea based Ready to Use Complementary Food Supplements (Active Comparator)
  Interventions: Dietary Supplement: Chick-pea based Ready to Use Complementary Food Supplements

INTERVENTIONS:
Dietary Supplement: Pushti packet — A food composed of roasted rice, roasted lentil, molasses and soybean oil
  Other Names: A food composed of roasted rice, roasted lentil, molasses and soybean oil
  Arms: Pushti Packet
Dietary Supplement: Rice based Ready to Use Complementary Food Supplements — A rice based diet.
  Arms: Rice based Ready to Use Complementary Food Supplements
Dietary Supplement: Chick-pea based Ready to Use Complementary Food Supplements — A chick-pea based diet.
  Arms: Chick-pea based Ready to Use Complementary Food Supplements

SUMMARY:
The prevention of malnutrition among children under 5 years of age requires consumption of nutritious food, including exclusive breast feeding for the first six months of life, followed by breastfeeding in combination with complementary foods thereafter until at least 24 months of age; a hygienic environment; access to preventive as well as curative health services, and good prenatal care. The proposed research is on the possible options for providing a nutritious diet, realizing the constraints of poverty and food insecurity faced by care givers whose children are at risk of developing or confirmed to be suffering from moderate malnutrition. Even when people are not typically food insecure but consume a relatively monotonous diet with few good-quality foods, they also have to have options for dietary improvement, and especially the possibility of ready-to-use complementary food supplements (RUCFS) for young children. This proposed research on development of RUCFS will pave the way for programmatic considerations for expansion of the use of new complementary food supplements for preventing malnutrition among young children in Bangladesh.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 18 months; either sex, having no acute illness, and be on at least one semi-solid or solid food in a day.

Exclusion Criteria:

* loss of appetite,
* oral lesion,
* congenital anomaly/acquired disorder affecting growth,
* severe acute malnutrition (SAM) defined by:

  * MUAC < 115 mm or
  * WL < -3 Z score or
  * bipedal edema,
  * persistent diarrhea,
  * tuberculosis,
  * any other chronic illness.

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Acceptability of at least one Ready -to-Use Complementary Food supplement | 7 days
  At least one of the experimental Ready -to-Use Complementary Food supplement will be acceptable to the study participants for prevention of malnutrition. The acceptability will be assessed by a 7-point Hedonic scale.

CONTACTS AND LOCATIONS:
Locations (1):
- ICDDR,B, Dhaka, Dhaka Division, Bangladesh

REFERENCES:
- [Derived] Ahmed T, Choudhury N, Hossain MI, Tangsuphoom N, Islam MM, de Pee S, Steiger G, Fuli R, Sarker SA, Parveen M, West KP Jr, Christian P. Development and acceptability testing of ready-to-use supplementary food made from locally available food ingredients in Bangladesh. BMC Pediatr. 2014 Jun 27;14:164. doi: 10.1186/1471-2431-14-164. PMID 24972632